CLINICAL TRIAL: NCT07321873
Title: A Phase 2b, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging Study to Evaluate the Efficacy and Safety of JNJ-88545223 For the Treatment of Participants With Active Psoriatic Arthritis
Brief Title: A Study to Evaluate the Efficacy and Safety of JNJ-88545223 for the Treatment of Participants With Active Psoriatic Arthritis
Acronym: VELOTA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 88545223PSA2001; 2025-523141-10-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2026-01-05; First posted 2026-01-07 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Arthritis, Psoriatic
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm 1: Placebo (Placebo Comparator): Participants will receive matching placebo to JNJ-88545223, from Week 0 to Week 16.
  Interventions: Drug: Placebo
- Arm 2: JNJ-88545223 Dose 1 (Experimental): Participants will receive JNJ-88545223 Dose 1 from Week 0 to Week 16.
  Interventions: Drug: JNJ-88545223
- Arm 3: JNJ-88545223 Dose 2 (Experimental): Participants will receive JNJ-88545223 Dose 2 from Week 0 to Week 16.
  Interventions: Drug: JNJ-88545223
- Arm 4: JNJ-88545223 Dose 3 (Experimental): Participants will receive JNJ-88545223 Dose 3 from Week 0 to Week 16.
  Interventions: Drug: JNJ-88545223

INTERVENTIONS:
Drug: JNJ-88545223 — JNJ-88545223 will be administered orally.
  Arms: Arm 2: JNJ-88545223 Dose 1; Arm 3: JNJ-88545223 Dose 2; Arm 4: JNJ-88545223 Dose 3
Drug: Placebo — Placebo will be administered orally.
  Arms: Arm 1: Placebo

SUMMARY:
The purpose of this study is to evaluate how well the study drug JNJ-88545223 works compared with a placebo (an inactive substance) in adults with active psoriatic arthritis (PsA). The study aims to see whether treatment with JNJ-88545223 can help reduce the signs and symptoms of PsA and improve joint and skin health.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of psoriatic arthritis (PsA) for at least 3 months before the first administration of study intervention and meet classification criteria for Psoriatic Arthritis (CASPAR) at screening
* Have active PsA as defined by: (a) At least 3 swollen joints and at least 3 tender joints at screening and at baseline (b) C-reactive protein (CRP) greater than or equal to (>=) 0.1 milligrams per deciliter (mg/dL) at screening from the central laboratory
* Have >= 1 of the following PsA subsets: distal interphalangeal joint involvement, polyarticular arthritis with absence of rheumatoid nodules, asymmetric peripheral arthritis, or spondylitis with peripheral arthritis
* Have active plaque psoriasis with at least one psoriatic plaque of >= 2 centimeter (cm) diameter or nail changes consistent with psoriasis
* A female participant of childbearing potential must have a negative highly sensitive serum pregnancy test (Beta-hCG) at screening and a negative urine pregnancy test at Week 0 prior to administration of study intervention

Exclusion Criteria:

* Has a nonplaque form of psoriasis (for example, erythrodermic, guttate, or pustular)
* Has a history or current signs or symptoms of severe, progressive, or uncontrolled renal, hepatic, cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic (except PsA), psychiatric, genitourinary, or metabolic disturbances
* Has suspected or known allergies, hypersensitivity, or intolerance to JNJ-88545223 or excipients used in the investigational medicinal product (IMP), including placebo (JNJ-88545223 investigator's brochure); or has a history of severe allergic reaction, angioedema, or anaphylaxis to drugs or food
* Has fibromyalgia or osteoarthritis symptoms that, in the opinion of the investigator, would have potential to interfere with efficacy assessments
* Currently has a malignancy or has a history of malignancy within 5 years prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2026-01-15 (Actual); Primary Completion 2027-06-28 (Estimated); Study Completion 2027-08-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants who Achieved an American College of Rheumatology (ACR) 50 Response at Week 16 | Week 16
  The ACR 50 responders are participants with an improvement of greater than or equal to (>=) 50 percent (%) from baseline in both the tender and swollen joint count and in at least 3 of the 5 assessments (patient's assessment of pain visual analog scale [VAS], patient's global assessment of disease activity [arthritis, VAS] scale, Physician's global assessment of disease activity VAS scale, Health Assessment Questionnaire and C-reactive protein).

SECONDARY OUTCOMES:
Proportion of Participants Who Achieved Psoriatic Area and Severity Index (PASI) 75 Response at Week 16 Among Participants with Baseline Body Surface Area (BSA) Greater Than or Equal to (>=) 3 Percent (%) and With Baseline IGA Score of >=2 | Week 16
  A PASI 75 response represents participants who achieved at least a 75 percent improvement from baseline in the PASI score. The PASI is a system used for assessing and grading the severity of psoriatic lesions. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas were assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 to 6, and for erythema, induration, and scaling, which are each rated on a scale of 0 to 4. The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease.
Proportion of Participants Who Achieved PASI 90 Response at Week 16 Among Participants with Baseline BSA >=3% and With Baseline IGA Score of >=2 | Week 16
  A PASI 90 response represents participants who achieved at least a 90 percent improvement from baseline in the PASI score. The PASI is a system used for assessing and grading the severity of psoriatic lesions. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas were assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 to 6, and for erythema, induration, and scaling, which are each rated on a scale of 0 to 4. The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease.
Proportion of Participants Who Achieved PASI 100 Response at Week 16 Among Participants with Baseline BSA >=3% and With Baseline IGA Score of >=2 | Week 16
  A PASI 100 response represents participants who achieved at least a 100 percent improvement from baseline in the PASI score. The PASI is a system used for assessing and grading the severity of psoriatic lesions. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas were assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 to 6, and for erythema, induration, and scaling, which are each rated on a scale of 0 to 4. The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease.
Proportion of Participants who Achieved an ACR 20 Response at Week 16 | Week 16
  The ACR 20 responders are participants with an improvement of >= 20% from baseline in both the tender and swollen joint count and in at least 3 of the 5 assessments (patient's assessment of pain VAS, patient's global assessment of disease activity [arthritis, VAS] scale, Physician's global assessment of disease activity VAS scale, Health Assessment Questionnaire and C-reactive protein).
Proportion of Participants who Achieved an ACR 70 Response at Week 16 | Week 16
  The ACR 70 responders are participants with an improvement of >= 70% from baseline in both the tender and swollen joint count and in at least 3 of the 5 assessments (patient's assessment of pain VAS, patient's global assessment of disease activity [arthritis, VAS] scale, Physician's global assessment of disease activity VAS scale, health assessment questionnaire and C-reactive protein).
Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) Score At Week 16 | Baseline up to Week 16
  The HAQ-DI score consists of questions referring to 8 categories: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and common daily activities. Responses in each functional area are scored from 0 to 3 (0=no difficulty and 3=inability to perform a task in that area). Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3 where 0 = least difficulty and 3 = extreme difficulty.
Change From Baseline in 36 Item Short Form Survey (SF-36) Physical Component Summary (PCS) Score at Week 16 | Baseline up to Week 16
  SF-36 is a standardized survey evaluating 8 aspects of functional health and wellbeing: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. The score for a domain was an average of the individual question scores, which were scaled 0 to 100 (100=highest level of functioning). Score from physical function, role physical, bodily pain, and general health domains were averaged to calculate PCS. Total score range for PCS was 0-100 (100=highest level of physical functioning).
Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to Week 16
  An AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product that does not necessarily have a causal relationship with the intervention. A SAE is any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a suspected transmission of any infectious agent via a medicinal product, and is medically important.
Number of Participants With Change from Baseline in the Laboratory Parameters | Baseline up to Week 16
  Participants with change from baseline in the laboratory parameters (hematology and serum chemistry) will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (4):
- United States (4):
  - Rheumatology Center of San Diego, San Diego, California
  - Joint and Muscle Research Institute, Charlotte, North Carolina
  - Paramount Medical Research & Consulting, Middleburg Heights, Ohio
  - Clinical Research Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency